CLINICAL TRIAL: NCT04099706
Title: Treatment of Chronic Postherpetic Pain With Autologous Fat Grafting - A Randomized Clinical Trial
Brief Title: Treatment of Chronic Postherpetic Pain With Autologous Fat Grafting - A RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Martin Sollie, Principal investigator, M.D, Dept. of Plastic and Reconstructive Surgery, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: S-20190112
Record Dates: First submitted 2019-08-27; First posted 2019-09-23 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Postherpetic Neuralgia; Shingles; Varicella Zoster; Herpes Zoster; Chronic Pain
Keywords: Chronic pain; Postherpetic Neuralgia
MeSH Terms: conditions — Neuralgia, Postherpetic; Herpes Zoster; Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The allocation will be masked. All patients will undergo the procedure under general anaesthesia. The randomized allocation will take place during surgery.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention - Fat grafting (Experimental): The participant will undergo the procedure under general anaesthesia. A small amount of fat (20-120 cc) will be harvested using liposuction, from the abdomen or the thighs. Randomized allocation will be made and when allocated to the intervention group, the fat will be purified using decanting and injected into the painful areas of skin.
  Interventions: Procedure: Autologous Fat Grafting / Fat Transplant
- Control - Saline (Sham Comparator): The participant will undergo the procedure under general anaesthesia. A small amount of fat (20-120 cc) will be harvested using liposuction, from the abdomen or the thighs. Randomized allocation will be made and when allocated to the control group, the fat will be discarded and saline will be injected into the painful areas of skin.
  Interventions: Procedure: Autologous Fat Grafting / Fat Transplant

INTERVENTIONS:
Procedure: Autologous Fat Grafting / Fat Transplant — See arm descriptions.

SUMMARY:
This randomized clinical trial investigates the possible beneficial effect of autologous fat grafting on postherpetic neuralgia.

DETAILED DESCRIPTION:
Herpes Zoster (HZ), is a condition caused by Varicella-Zoster virus (VZV), The disease is caused by reactivation of a latent VZV-infection in the sensory ganglia.

Clinically the condition is characterized by a painful, unilateral, vesicular rash. Pain is the most prominent symptom in around 90% of patients. In 10% of patients, this pain remains and becomes chronic.

Post-herpetic neuralgia is a chronic pain syndrome that occurs after the dermal manifestation disappears. Treatment is complex and mainly topical or systemic. For many patients, this is not sufficient and they live with constant pain.

Autologous fat grafting has shown promise in treating several different painful conditions such as post-mastectomy pain syndrome, painful scars, etc. Our previous pilot study (NCT03584061) investigating the effect of autologous fat grafting on PHN, showed a marked reduction in pain with half of the patients being pain-free after the procedure.

The aim of this study is to test the hypothesis that autologous fat grafting is more effective than a sham operation in treating PHN.

ELIGIBILITY:
* Inclusion Criteria:
* Age over 18
* Pain in area of former VZV-infection.
* Pain present over 3 months after reactivation of VZV and is present at least 4 days a week and of intensity >3 on the VAS-scale
* Exclusion criteria:
* Psychiatric illness that could potentially affect the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-09-19 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Neuropathic pain [LEVEL OF PAIN] | 6 months
  Neuropathic Pain Symptom inventory (NPSI), Questionnaire. NPSI consists of 12 items in total: 10 items investigates differential symptoms descriptors and 2 items evaluate spontaneous and paroxysmal spontaneous pain.
  The tool evaluates mean pain intensity in the last 24h in a verbal numeric scale from zero (no pain) to 10 (worst imaginable pain). Total pain intensity score may be calculated by the sum of the 10 descriptors.
  The descriptors are:
  Burning, Squeezing, Pressure, Electric Shocks, Stabbing, Provoked by brushing. Provoked by pressure, Evoked by cold stimulation, Pins and needles, Tingling.

SECONDARY OUTCOMES:
Quality of life [QUALITY OF LIFE/ SATISFACTION] | 6 months
  Short Form 36 (SF-36), Questionnaire. Scoring the RAND 36-Item Health Survey is a two-step process. First, precoded numeric values are recoded per a scoring key. All items are scored so that a high score defines a more favorable health state. Each item is scored on a 0 to 100 range so that the lowest and highest possible scores are 0 and 100, respectively. Scores represent the percentage of total possible score achieved. After this, items in the same scale are averaged together to create the 8 scale scores.
  The eight health concepts are: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. It also includes a single item that provides an indication of perceived change in health.

CONTACTS AND LOCATIONS:
Overall Officials: Jens Ahm Sorensen, Prof, Principal Investigator — Professor
Locations (1):
- Odense University Hospital, Odense, Funen, Denmark

IPD SHARING:
Plan to Share IPD: No